CLINICAL TRIAL: NCT01095718
Title: Comparison of 3 Learning Methods and Their Underlying Mechanisms to Improve Independent Living in the Activities of Daily Living in Alzheimer's Dementia: a Randomized Controlled Trial
Brief Title: Comparison of 3 Learning Methods to Improve Independent Activities of Daily Living (IADLs) in Alzheimer Disease
Acronym: C3LM-ILAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Clinical Research and Innovation (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Fondation Mederic Alzheimer (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Department of Clinical research and innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ID RCB 2009-A01303-54
Record Dates: First submitted 2010-03-15; First posted 2010-03-30 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2011-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Errorless Learning (Experimental): Errorless learning refers to the use of feedforward instruction before actions to prevent learners from making mistakes. The therapist presents steps with the following instruction and the visual cues e.g., Here are steps that you need to do to make some coffee, please repeat them".
  The therapist gives cues before the completion of each step. At each step the patient receives verbal and visual cues. Then cue cards are hidden, and the therapist asks immediately to give the answer about the step involved.
  The therapist allows the participant to try finding the solution, if the answer or action is not immediately given, the participant receives a cue, and moves to the next step.
  During cueing the patient will mostly receive verbal and visual cues and if necessary physical help.
  Interventions: Behavioral: Errorless Learning
- Modeling (Active Comparator): The therapist gives the same tailored baseline information for each task. The therapist issue specific information for each step.Using tailored mastery modeling, the therapist shows the steps in front of the patient. There is a special emphasis on adjusting the modeling just above the patient's abilities.
  The therapist does the steps, at the same time he/she uses verbal cues during the performance. Then the therapist asks immediately to the patient to do the steps.
  Interventions: Behavioral: Modeling
- Trial and Error (Active Comparator): Trial and Error refers to the regular unstructured learning and is considered as control condition.
  Here the patient is encouraged to complete the task. When there is mistake, the therapist corrects it. Verbal cues will only be provided if the patient is unable to find and complete the correct next step or commit mistakes. The therapist use general instruction: "Here is "task", I will ask you to "actions"", followed by specific instruction, "and I will help you after you have tried".
  Interventions: Behavioral: Trial and Error

INTERVENTIONS:
Behavioral: Errorless Learning — Errorless learning refers to the use of feedforward instruction before actions to prevent learners from making mistakes. The therapist presents steps with the following instruction and the visual cues e.g., Here are steps that you need to do to make some coffee, please repeat them".
  The therapist gives cues before the completion of each step. At each step the patient receives verbal and visual cues. Then cue cards are hidden, and the therapist asks immediately to give the answer about the step involved.
  The therapist allows the participant to try finding the solution, if the answer or action is not immediately given, the participant receives a cue, and moves to the next step.
  During cueing the patient will mostly receive verbal and visual cues and if necessary physical help.
  Arms: Errorless Learning
Behavioral: Modeling — The therapist gives the same tailored baseline information for each task. The therapist issue specific information for each step. Using tailored mastery modeling, the therapist shows the steps in front of the patient. There is a special emphasis on adjusting the modeling just above the patient's abilities.
  The therapist does the steps, at the same time he/she uses verbal cues during the performance.
  Then the therapist asks immediately to the patient to do the steps.
  Arms: Modeling
Behavioral: Trial and Error — The therapist gives the same tailored baseline information for each task. The therapist issue specific information for each step. Using tailored mastery modeling, the therapist shows the steps in front of the patient. There is a special emphasis on adjusting the modeling just above the patient's abilities.
  The therapist does the steps, at the same time he/she uses verbal cues during the performance.
  Then the therapist asks immediately to the patient to do the steps.
  Arms: Trial and Error

SUMMARY:
This study is a comparison of 3 learning techniques, Errorless learning, modelling and trial and error, in the relearning of IADL of Alzheimer patients from mild to moderately severe dementia.

Tailored IADL will be chosen for each patient (n=300) and trained in individualized sessions for 6 weeks.

This study focuses on the relationship between learning techniques, IADL and memory processes, in a threefold way:

1. it will determine which of the of the three learning techniques (EL, MR, TE) will improve most the (re)learning of instrumental skills in different dementia stages using a randomized controlled trial;
2. it will explain the role of implicit and explicit memory mechanisms in the (re)learning of IADL tasks; and
3. as a secondary objective, it will explore the possible drug treatment by behavioral intervention interaction effects of the three learning techniques.

DETAILED DESCRIPTION:
Scientific background and rationale Alzheimer dementia (AD) is the most common cause of progressive cognitive deterioration that alters memory and learning to such a degree that it heavily interferes with daily living. Functional autonomy loss is a key feature of AD, as it follows a slow degradation process in cognitive function and in the ability to perform instrumental activities of daily living (IADL), such as managing finance, food preparation or using a dish washer. Normally, learning occurs in an unstructured manner, which consists of guessing and the occurrence of errors during acquisition (Trial and Error, TE). However, there is abundant evidence that reducing errors during learning (Errorless Learning, EL) or increasing the time period between recall attempts (Modeling with Spaced Retrieval, MR) allow even moderate and severe Alzheimer Dementia (AD) patients to (re)learn instrumental activities of daily living (IADL) such as using a new route, an agenda or a cassette/radio player. While these findings are encouraging, we still do not fully understand the memory mechanisms underlying different learning techniques that are crucial in improving IADL tasks (re)learning and remembering in AD patients. Because acetyl cholinesterase inhibitors or memantine may be active moderators of intervention targeting memory improvement, complex intervention using behavioral enrichment training should explore any drug treatment by behavioral intervention interaction effects.

Description of the project methodology

This study focuses on the relationship between learning techniques, IADL and memory processes, in a threefold way:

1. it will determine which of the of the three learning techniques (EL, SR, TE) will improve most the (re)learning of instrumental skills in different dementia stages using a randomized controlled trial;
2. it will explain the role of implicit and explicit memory mechanisms in the (re)learning of IADL tasks.; and
3. it will explore the possible drug treatment by behavioral intervention interaction effects of the three learning techniques.

   * Primary outcome :

Is the (re)learning effectiveness (physical performance) of each procedure and the overall maintain of the autonomy. All intervention are individualized training. The learning procedure comparison will allow us to assess the (re) learning capacities of IADL tasks in AD patients according to severity stages from mild to moderately severe.

• Secondary outcome : Assessing the role of the implicit memory processes over the explicit memory processes in the (re)learning of IADL tasks. Overall effects of the intervention over the patient's autonomy, cognitive functioning, behavioral disturbances, quality of life and careers burden.

Settings: Nursing Homes, Day Care centers, Memory Clinics Locations: Nijmegen, The Netherlands and Nice and Bordeaux agglomerations, France 3 different interventions given in individual sessions at participant's facility.

Each intervention is a 6-week training with a post assessment at 4-week follow-up. Each participant will receive one of the 3 interventions for 2 hours twice a week in individual sessions.

Errorless learning(EL) refers to the use of feedforward instruction (i.e., how to do) before actions to prevent learners from making mistakes.

Modeling with Spaced Retrieval (MR) techniques refers to the modeling of the steps and the increasing time interval between the completion of the task and the rehearsal of the targeted information by the patient.

Trial and Error (TE) refers to the regular unstructured learning and is considered as control condition.

A standardized 1-week training has been developed in French and Dutch to train French and Dutch therapists at each learning techniques.

ELIGIBILITY:
Inclusion criteria:

* Having a diagnosis of mild to moderately severe Alzheimer Dementia type with a MMSE score between 10 and 26;
* Fulfill the DSM-IV-TR and NINCDS-ADRDA criteria for Alzheimer's dementia type (33;34);
* Aged 60 and older;
* Not able to complete without cue the proposed tasks during the screening interview.
* Having a Social Security System

Exclusion criteria:

* MMSE < 10 or > 26
* Participants with severe deficits in alertness,
* Deemed behavioral disturbances (e.g., such as high NPI irritability symptom as defined with a score of 6 or above out of a maximum score of 12),
* Known medications that could interfere with the intervention (except AD medication, cf AD treatments).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the intervention will be the performance and errors of participants. Each task is comparable as the assessment procedure remains the same across disease stages. | 2 hours - 2 times a week during 6 weeks

SECONDARY OUTCOMES:
Baseline neuropsychological assessments. Premorbid intelligence level will be estimated by the National Adult Reading Test (NART). The Mini Mental State Examination (MMSE) will be used to assessed cognitive status. | 3 times through the trial

CONTACTS AND LOCATIONS:
Overall Officials: Robert Philippe, MD, PhD, Principal Investigator — Centre Mémoire CHU de Nice
Locations (1):
- CHU de Nice Centre Mémoire, Nice, France